CLINICAL TRIAL: NCT06156176
Title: Pursuing Reduction in Fatigue After COVID-19 Via Exercise and Rehabilitation (PREFACER): A Randomized Feasibility Trial
Acronym: PREFACER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lawson Research Institute of St. Joseph's (Other)
Collaborators: Western University, Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PBPREFACER01
Record Dates: First submitted 2023-10-30; First posted 2023-12-05 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-04

CONDITIONS: Long-COVID; Long COVID-19; Post-COVID-19 Syndrome; Post-COVID Syndrome; Fatigue; Post COVID-19 Condition; Post-COVID Condition
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue

STUDY DESIGN:
Intervention Model Description: There are two parallel treatment groups: COVIDEx rehabilitation program and standard of care.
Who Masked: Outcomes Assessor
Masking Description: Outcome Assessors (physiotherapists) will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVIDEx (Experimental): This group will receive two 50-minute rehabilitation sessions per week for 8 weeks.
  Interventions: Other: COVIDEx
- Standard of Care (No Intervention): This group will receive standard of care (no intervention) for the 8-week intervention period.

INTERVENTIONS:
Other: COVIDEx — The COVIDEx intervention was developed by triangulating patient preferences/needs, clinicians' expertise, and best current evidence specific to Long COVID and adapted from interventions for other complex fatigue disorders, which are consistent with evidence informed practice. The program is delivered by trained instructors and comprises of two 50-minute sessions each week for eight weeks. The intervention is designed to be delivered virtually in groups of 6 patients, to eliminate travel requirements for the study. The components of the program are: (i) warm-up (1 min), (ii) cardio training (5 min), (iii) rest (3 min), (iv) balance training (5 min), (v) breathing exercises (3 min), (vi) cognitive training (5 min), (vii) strengthening training (5 min), and (viii) stretching (10min). The COVIDEx program will be paced in order to prevent post-exertional malaise (PEM) in participants.
  Arms: COVIDEx

SUMMARY:
Long COVID is a complex condition that affects approximately 1.4 million Canadians following SARS-CoV-2 infection. Fatigue is the most common symptom of Long COVID. This feasibility trial will evaluate a new rehabilitation program called COVIDEx for treating fatigue after COVID-19, and compare its effectiveness to the standard treatment currently used. The experimental treatment group will receive an 8-week multi-modal rehabilitation program with two 50-minute sessions per week. 60 participants will be recruited, randomly assigned to the COVIDEx program or standard of care (SoC) and followed for 24 weeks.

DETAILED DESCRIPTION:
The investigators propose a modified Zelen, randomized, single-centre, feasibility trial with two parallel groups (intervention vs standard of care). Zelen designs are recommended for evaluating interventions - specifically, to estimate effectiveness rather than efficacy - under real-world conditions of incomplete adherence. Thus, the proposed design is particularly well suited to examine rehabilitation interventions for Long COVID. Participants will be identified and recruited from the community and St. Joseph's Post-Acute COVID-19 outpatient program at Parkwood Institute. Once the clinician and research personnel have determined eligibility, they will log into the web-based computer-generated randomization system. The randomization scheme will be constructed using varying, permuted blocks, stratified by sex and hospitalized status (1 = hospitalized, 0 = otherwise). In alignment with the modified Zelen design's unique approach, all participants will be randomized before obtaining their informed consent. However, immediately after randomization, all participants, irrespective of their group, will be informed and asked to consent to the following:

All participants will be informed that they are part of an observational study designed to follow the natural progression of Long COVID and to evaluate the costs associated with standard post-COVID-19 treatments. This includes both the COVIDEx and SoC groups. The objective is to ensure comprehensive data collection on health outcomes and healthcare utilization across the spectrum of post-COVID care. By blinding patients to the presence of the experimental group, the modified Zelen design will mitigate the effects of feeling disappointed, frustrated, or discouraged about being assigned SoC, which is important given the primary outcome is a subjective, patient reported outcome measure (detection bias). This approach will also reduce the likelihood that patients in the SoC group begin self-motivated programs trying to mimic the intervention (performance bias) since there is no standard of care for this population. Upon completion of the study, both groups will attend a disclosure interview where the randomized nature of the study will be revealed, the rationale for this deception/treatment delay will be provided and full informed consent to use their data for the RCT will be sought. The deception disclosure interview for participants will occur over the phone. A member of the Parkwood research team (research coordinator or research assistant) will telephone each control group participant upon completion of the participant's study procedures and disclose the deception to participants. While on the phone, a copy of the debriefing letter of information/consent (LOI/C) will be emailed to the participant, for the participant to read. The research coordinator or assistant will answer any questions that the participant has and give the participant as much time is needed to sign the consent form. SoC patients will then be offered the COVIDEx intervention. The treatment period will be 8 weeks, with 2 COVIDEx sessions per week.

Outcomes will be collected at baseline, 4-, 8-, 12- and 24- weeks follow-up during assessment sessions. Outcomes include feasibility measures and clinical outcomes, including a transcranial magnetic stimulation (TMS) brain function test. Qualitative one-on-one interviews will explore the acceptability of the intervention and barriers/facilitators to intervention adherence and study retention. Only participants randomized to the COVIDEx group will be asked to participate in the interviews. The study team will not gather data from control group participants if they choose to participate in the COVIDEx intervention.

Measurement of post-exertional malaise (PEM): Some participants may indicate that they experience PEM on the demographic questionnaire. PEM is defined as the worsening of symptoms (such as difficulty thinking, problems sleeping, sore throat, headaches, feeling dizzy, or severe tiredness) after a physical or mental activity that would not have caused a problem before COVID-19 infection and subsequent post-COVID-19 fatigue. We will address this in the trial by: (1) Pacing the COVIDEx session to prevent over-exertion. A pacing strategy and protocol may reduce exacerbation of PEM for those with Long COVID. Pacing will entail frequently gathering subjective measurements of intensity from participants, as well as ensuring that all components of the session (i.e., cardio, strength training) have adequate rest and recovery in between periods of more intense activity. Participants will inform the physiotherapist or exercise instructor of their resting heart rate and blood oxygen levels before each session and after each component of the session, which will help determine exercise intensity and pacing. (2) Monitoring blood lactate levels in participants. All COVIDEx participants, throughout the COVIDEx sessions, will use an Apple Watch to monitor surrogate measures for their blood lactate levels (specifically, heart rate, blood oxygen, steps activity, and sleep). This device is required to be worn by participants as often as possible over the 24-week study period, but especially during each COVIDEx session. Monitoring surrogate measures for blood lactate enables examination of metabolic responses (i.e., mitochondrial dysfunction, reduced tissue oxygenation) in individuals with Long COVID, which could help prevent the onset of PEM by ensuring participants do not exceed a threshold that could induce PEM. Specifically, our objective of monitoring surrogate measures for blood lactate is for safety purposes to prevent overreaching in participants with Long COVID. Participants will be asked to inform the physiotherapist or exercise professional of their blood oxygen levels and heart rate at various time points throughout the COVIDEx intervention, so the instructor can gauge intensity and modify exercise intensity as needed. The instructor will have a lactate range table on hand to ensure participants are within the Safe and Functional Overreaching zones (stated within the research plan) and will approximate this based on participant's blood oxygen levels. The Apple Watches will be provided to participants at no cost to them. Participants have the choice to use their own Apple Watch or can be provided one from the study team. Participants may be required to input basic profile information on the wearable device, such as email, age, height, weight, and/or gender to personalize the tracking features.

To also assist in assessing PEM and fatigue, an ecological momentary assessment (EMA) design will be used to ask participants how they're feeling at random time-points after participating in the COVIDEx sessions (up to the 24-week follow-up). For comparison, participants in the control group will also be administered the EMA questions. These questions are based off the DePaul Symptom Questionnaire-SF. Participants will be asked to download the ExpiWell app, which will be the way of administering the questions at random time-points. Collecting EMA data will assist the researchers in identifying potential cases of PEM and/or any other adverse or serious adverse events. EMA data will be collected for 24 weeks once the participant signs the LOI and agrees to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults of at least 18 years of age
* Able to provide informed consent
* Can speak and understand English
* Documented history of SARS-CoV-2 infection (positive PCR/antigen test during acute illness or clinical diagnosis by physician during or after the acute illness)
* Fatigue symptoms within 3 months of COVID-19 infection, lasting at least 2 months
* Fatigue symptoms cannot be explained by an alternative diagnosis
* Fatigue symptoms may be new onset following initial recovery from an acute COVID-19 infection or persist from the initial illness
* Fatigue symptoms may have an episodic nature, fluctuate or relapse over time
* Minimal functional capability: able to walk 10-15 minutes and be recovered within 30-60 minutes or without significant post-exertional malaise (PEM)
* Has applicable technology to access Microsoft Teams and Webex (i.e., computer, laptop, tablet)

Exclusion Criteria:

* Active SARS-CoV-2 infection
* Pre-existing physical, cognitive, and/or mental health conditions that make exercise contraindicated, consent unattainable, or that cause symptoms similar to those seen in post COVID-19 (e.g., major neurocognitive disorder, schizophrenia, chronic fatigue syndrome) that could affect data
* Inability to follow study procedures
* Pregnant and/or breastfeeding
* Received investigational agents as part of a separate study within 30 days of the screening visit
* Has any type of metal bodily implant in head or heart (i.e., pins, plates, pacemakers)
* Current participation in other studies related to COVID-19, exercise, and/or fatigue interventions OR participation within 30 days of the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment | Baseline
  The number of screened patients who are eligible, the proportion of eligible patients who consent, number of patients enrolled per month, reasons for non-enrolment.
Intervention Fidelity | Week 24
  The proportion of participants who meet the acceptable level of intervention fidelity (>80%). A fidelity checklist will be used to assess feasibility that includes adherence (i.e., delivery of each key component of the intervention-absent/present), dosage (amount of intervention delivered, number of sessions completed, overall duration of sessions), quality of intervention delivery (i.e., mode of delivery of COVIDEx), and participant acceptability (extent to which participants in the intervention group found the intervention useful).
Retention | Week 24
  The proportion of missed assessments and incomplete outcome measures data, and proportion of participants who withdraw from the trial.
Zelen Design Acceptability | Week 24
  The proportion of patients in the standard of care group who provide consent to include their data in the RCT following the disclosure interview.

SECONDARY OUTCOMES:
Change in 30-Second Sit-to-Stand Test | Baseline to Week 24
  The 30-Second Sit-to-Stand Test involves repeatedly standing up from and sitting down on a chair within a 30-second time frame, assessing lower body strength and functional fitness in individuals. Participants are timed for 30 seconds and the number of times they stand up and sit down in a chair in the 30-second period is recorded. More repetitions indicate higher functional ability (i.e., endurance, leg strength).
Change in Borg Scale of Perceived Physical Exertion | Baseline to Week 24
  The Borg Rating of Perceived Exertion (RPE) is a subjective scale used to assess an individual's perceived intensity of physical activity, providing a measure of their effort level during exercise. We are using the 6-20 scale (6 being easy exercise to 20 being extremely vigorous). Participants rate how difficult exercise/activity feels from 6 (no exertion at all) to 20 (maximal exertion).
Change in The DePaul Symptom Questionnaire | Baseline to Week 24
  The DePaul Symptom Questionnaire (DSQ) is a self-report instrument used to assess the severity and frequency of symptoms related to chronic fatigue syndrome in individuals, covering various domains including fatigue, sleep, and cognitive issues. Participants' physical symptoms are rated on a five-point scale for frequency (0=none of the time, to 4=all of the time) and severity (0=no symptoms, 4=very severe).
Change in DePaul Symptom Questionnaire - Post-Exertional Malaise (short-form) | Baseline to Week 24
  Post-Exertional Malaise (PEM) will be assessed using the DSQ-PEM-SF. This questionnaire is used to assess the severity and frequency of symptoms related to PEM in individuals, covering various domains including fatigue, sleep, and cognitive issues.
Change in EQ-5D-5L | Baseline to Week 24
  The EuroQol 5 Dimension 5 Level (EQ-5D-5L) is a standardized, self-reported, health-related quality of life questionnaire that assesses individuals across five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) with three levels of severity ("no problems" to "extreme problems"), providing a simple and widely used measure for health outcome assessments.
Change in Global Rating of Change Scale | Baseline to Week 24
  The GRoC (Global Rating of Change Scale) Scale is a tool designed to assess individuals' subjective perceptions of change over time, typically used to measure the effectiveness of interventions or treatments by comparing current status to a previous baseline. Participants will rate the change in their symptoms from -5 (much worse) to +5 (much better) and we'll be assessing change in post-COVID fatigue.
Change in Hospital Anxiety and Depression Scale | Baseline to Week 24
  The Hospital Anxiety and Depression Scale (HADS) is a self-report questionnaire designed to assess and measure the levels of anxiety and depression in individuals. Statements are rated on a scale of 0 to 3 for how true they are for the participant. A higher score indicates a worse outcome (anxiety or depression).
Change in Post-COVID-19 Functional Status | Baseline to Week 24
  This form will collect information on a person's abilities to perform daily activities (and any limitations such as symptoms, pain, or depression). Effect of COVID-19 on functional status is graded on a 5-point scale from 0 (no functional limitations) to 4 (severe functional limitations).
Change in Fatigue | Baseline to Week 24
  The PROMIS (Patient-Reported Outcomes Measurement Information System) fatigue scale (short-form) is a self-report measure designed to assess the impact and severity of fatigue experienced by individuals. This scale will be used to measure participants' fatigue levels on a 5-point Likert scale at baseline and at weeks 4, 8, 12, and 24.
Change in Pain | Baseline to Week 24
  The Visual Analogue Pain Scale (VAS-Pain) is a subjective pain assessment tool where individuals mark their perceived pain intensity on a continuous line, that will range from "no pain" to "worst pain imaginable," providing a quick and visual measure of pain severity. Participants' pain levels will be measured at baseline, and at weeks 4, 8, 12, and 24.
Blinding Success Rate | Week 24
  Success rate of blinding of the outcome assessors will be evaluated with the James Blinding Index (JBI) scale. The JBI is a continuous value such that 0 <= James BI <= 1. If the index is 1, all responses are incorrect, and complete blinding is inferred, albeit this may indicate unblinding in the opposite direction (e.g. opposite guessing). If the index is 0, all responses are correct, and complete unblinding is inferred. If the index is 0.5, then half of the guesses are correct and half of the guesses are incorrect, inferring random guessing. Unblinding may be claimed if the upper limit of the two-sided confidence interval is < 0.5. The JBI will be evaluated at the end of the trial (24-weeks). A very short questionnaire will ask participants which group they thought they were in (COVIDEx or control, to assess the success of the blinding).
Change in Brain Function | Baseline to Week 24
  Brain function will be assessed using a Magstim Rapid II TMS system to measure Motor Evoked Potential amplitudes and cortical silent period durations of the first dorsal interosseous muscle and the tibialis anterior muscle in the dominant hemisphere's primary motor cortex using a 70 mm figure eight coil and 120mm V coil, respectively.
Burden of Outcome Measures Completeness | Week 24
  Proportion of missing visits, missing outcomes/data, and reasons for missingness.
Patient Perceptions | Week 24
  We will conduct one-on-one interviews with COVIDEx participants and treating physiotherapists at the end of the study protocol, to understand the acceptability of the intervention, perceived benefits, barriers/facilitators to adherence, implementation challenges, and experiences with the modified Zelen design. This will inform the extent to which it is feasible in a real-world setting. Participants will be asked to share their perspectives around study participation and completion to optimize our recruitment and retention strategies for the definitive trial.

CONTACTS AND LOCATIONS:
Overall Officials: Pavlos Bobos, PhD, Principal Investigator — Western University
Locations (1):
- Parkwood Hospital - St. Joseph's Health Care London, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pouliopoulou DV, Macdermid JC, Saunders E, Peters S, Brunton L, Miller E, Quinn KL, Pereira TV, Bobos P. Rehabilitation Interventions for Physical Capacity and Quality of Life in Adults With Post-COVID-19 Condition: A Systematic Review and Meta-Analysis. JAMA Netw Open. 2023 Sep 5;6(9):e2333838. doi: 10.1001/jamanetworkopen.2023.33838. PMID 37725376
- [Background] Pouliopoulou DV, Billias N, MacDermid JC, Miller E, O'Brien KK, Quinn KL, Malvankar-Mehta MS, Pereira TV, Cheung AM, Razak F, Stranges S, Bobos P. Prevalence of post-acute sequelae of SARS-CoV-2 infection in people living with HIV: a systematic review with meta-analysis. EClinicalMedicine. 2024 Dec 17;79:102993. doi: 10.1016/j.eclinm.2024.102993. eCollection 2025 Jan. PMID 39802304
- [Background] Pouliopoulou DV, Hawthorne M, MacDermid JC, Billias N, Miller E, Quinn K, Decary S, Razak FA, Cheung A, Galiatsatos P, Pereira TV, Bobos P. Prevalence and Impact of Postexertional Malaise on Recovery in Adults With Post-COVID-19 Condition: A Systematic Review With Meta-analysis. Arch Phys Med Rehabil. 2025 Aug;106(8):1267-1278. doi: 10.1016/j.apmr.2025.01.471. Epub 2025 Feb 5. PMID 39921187
- [Background] Saunders EG, Pouliopoulou DV, Miller E, Billias N, MacDermid JC, Brunton L, Pereira TV, Quinn KL, Bobos P. Rehabilitation interventions and outcomes for post-COVID condition: a scoping review. BMJ Public Health. 2025 Feb 26;3(1):e001827. doi: 10.1136/bmjph-2024-001827. eCollection 2025. PMID 40017924
- [Derived] Billias N, Pouliopoulou DV, Lawson A, D'Alessandro V, Bryant DM, Peters S, Rushton AB, Miller E, Brunton L, McGuire S, Nicholson M, Birmingham TB, MacDermid JC, Quinn KL, Razak F, Goulding S, Galiatsatos P, Saunders E, Marsh J, Pereira TV, Bobos P. Pursuing Reduction in Fatigue After COVID-19 via Exercise and Rehabilitation (PREFACER): a protocol for a randomised feasibility trial. BMJ Open. 2025 Nov 9;15(11):e102112. doi: 10.1136/bmjopen-2025-102112. PMID 41213692